CLINICAL TRIAL: NCT03042143
Title: Repair of Acute Respiratory Distress Syndrome by Stromal Cell Administration (REALIST): An Open Label Dose Escalation Phase 1 Trial Followed by a Randomised, Double-blind, Allocation Concealed, Placebo-controlled Trial.
Brief Title: Repair of Acute Respiratory Distress Syndrome by Stromal Cell Administration (REALIST)
Acronym: REALIST
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other); Northern Ireland Clinical Trials Unit (Other); NHS Blood and Transplant (Other Government)
Responsible Party: Principal Investigator, Professor Danny McAuley, Professor and Consultant of Intensive Care Medicine, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16154DMcA-AS
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome; Human umbilical cord-derived mesenchymal stem cells; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Plasma-lyte 148

STUDY DESIGN:
Intervention Model Description: The phase 1 trial is an open label dose escalation pilot study in which cohorts of subjects with moderate to severe ARDS will receive increasing doses of a single infusion of Realist Orbcel-C in a 3+3 design. Initially 3 cohorts with 3 subjects/cohort.
  In the completed Phase 1 REALIST trial, infusion of 400 million cells was achieved without any dose limiting toxicity at day 7 and has been approved by the DMEC as the intervention dose for this study.
  The phase 2 trial is a randomised, double-blind, allocation concealed placebo-controlled study using the maximal tolerable dose as determined by the DMEC in patients with moderate to severe ARDS due to COVID-19 or other causes of ARDS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The cell therapy facility and clinical trials pharmacist will be unblinded. The unblinded individuals will keep the treatment information confidential and will not discuss or release information on treatment allocation to the patient, the investigator, or other unauthorised personnel.
  As in prior studies of MSCs, the infusion bag containing either the cell product or placebo will be masked at the time of preparation in the clinical site's cell therapy facility so that the contents of the infusion bag are not visible to the investigators or to the clinicians who are administering the study drug. The contents of the infusion bag will be administered through a masked infusion set.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human umbilical cord derived CD362 enriched MSCs (Experimental): Maximum tolerated dose from the phase 1 trial will be infused over 30 to 90 mins
  Interventions: Biological: Human umbilical cord derived CD362 enriched MSCs
- Placebo (Plasma-Lyte 148) infusion (Placebo Comparator): Plasma-Lyte 148 infused over 30 to 90 mins
  Interventions: Biological: Placebo (Plasma-Lyte 148)

INTERVENTIONS:
Biological: Human umbilical cord derived CD362 enriched MSCs — Infusion of Human umbilical cord derived CD362 enriched MSCs
  Arms: Human umbilical cord derived CD362 enriched MSCs
Biological: Placebo (Plasma-Lyte 148) — Infusion of placebo
  Arms: Placebo (Plasma-Lyte 148) infusion

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) causes the lungs to fail due to the collection of fluid in the lungs (pulmonary oedema). ARDS is common in severely ill patients in Intensive Care Units and is associated with a high mortality and a high morbidity in those who survive. ARDS occurs in approximately 20% case of COVID-19 and respiratory failure is the leading cause of mortality. There is a large economic burden with direct healthcare costs, but also indirectly due to the impact on the carer and patient through the patients inability to return to full time employment. There is little evidence for effective drug (pharmacological) treatment for ARDS. There is increasing information that mesenchymal stem cells (MSCs) might be important in treating ARDS. REALIST will investigate if a single infusion of MSCs will help in the treatment of ARDS. The first step will be to first of all determine what dose of MSCs is safe and then divide patients suffering from ARDS into two groups, one of which will get MSCs and the other a harmless dummy (or placebo) infusion, who will then be followed up to determine if lung function improves. If effective this may lead to further research to determine if MSCs are effective in patients with ARDS.

DETAILED DESCRIPTION:
The role of MSCs as a novel treatment in ARDS. Mesenchymal Stem Cells (MSCs) are a mononuclear cell population that have the potential to differentiate into multiple lineages, and bone, cartilage and adipocyte cells in particular. Cell-based therapies have been termed the "next pillar of Medicine". MSCs constitute an innovative approach with substantial therapeutic promise for ARDS. MSCs possess several favorable biological characteristics, including convenient isolation, ease of expansion in culture while maintaining genetic stability, minimal immunogenicity and feasibility for allogenic transplantation.

MSCs reduce inflammation and enhance bacterial clearance during rodent and murine bacterial pneumonia, and augment repair of the animal and human lung. Large animal studies have also replicated these beneficial effects. Bone marrow derived (BM) hMSCs decreased acute lung injury (ALI), without producing organ toxicity, in endotoxin injured pigs. Two randomised small phase 1 studies of plastic adherent MSCs in patients with ARDS have taken place. In Japan, investigators used adipose-derived plastic adherent cells in a small cohort (n=12) of patients with ARDS randomized 1:1 to MSCs or placebo: showing that the cells were safe and well-tolerated in this patient group, and were associated with reduced plasma levels of the alveolar epithelial cell injury marker SP-D. In the US Matthay has completed the phase 1 START trial, using a dose escalation study of plastic adherent bone marrow derived MSCs, in patients with moderate to severe ARDS. START showed that marrow derived MSCs at similar doses to those proposed in this study are safe and well-tolerated, (n=9), with a trend to reduced lung injury in the group treated with the highest (10x10^6cells/kg) compared with the lower doses, 1-5x10^6cells/kg.

Current (20 March 2020) data on novel coronavirus disease (COVID-19) suggests that it causes a mortality rate of ~3.4%, compared with <0.1% with seasonal influenza. ARDS occurs in approximatel 20% cases of COVID-19 and respiratory failure is the leading cause of mortality. In a restropective multi-centre study of 150 confirmed cases in Wuhan, China, ARDS occured in significantly greater proportion of non-survivors 81% (55/68 patients) compared with only 9% survivors (7/82 patients); p<0.01. In another study of 193 confirmed COVID-19 cases, ARDS was observed at a significantly higher rate in non-survivors 93% (50/54 patients) compared with survivors, 7% (9/137) patients; p<0.0001.

During the current COVID-19 pandemic, MSCs have been administered in a pilot study of seven patients with COVID-19 pneumonia. A single infusion of 1 x 10^6 MSCs were administered intravenously when their condition was considered to be deteriorating despite other treatments, however only 1 of the 7 patients required critical care and mechanical ventilation. 4 patients were described as severe with compromise of respiratory function. Patients underwent follow up for 14 days and no infusional toxicity or adverse events were reported.

Trial design:

The phase 1 trial is an open label dose escalation pilot study in which cohorts of subjects with moderate to severe ARDS will receive increasing doses of a single infusion of Realist Orbcel-C in a 3+3 design. We initially plan 3 cohorts with 3 subjects/cohort. Planned doses for the 3 cohorts pending absence of safety concerns are 100 x 10^6 cells, 200 x 10^6 cells and 400 x 10^6 cells.

In the completed Phase 1 REALIST trial, infusion of 400 million cells was achieved without any dose limiting toxicity at day 7 and has been approved by the DMEC as the intervention for this study.

The phase 2 trial is a randomized, double-blind, allocation concealed placebo-controlled study using the 400x10^6 cell dose of Realist Orbcel-C in patients with moderate to severe ARDS due to either COVID-19 or other causes of ARDS.

Primary objective:

To assess the safety of a single intravenous infusion of MSCs in patients with ARDS due to either COVID-19 or other cause of ARDS.

Secondary objectives:

In patients with moderate to severe ARDS to determine the effect of a single intravenous infusion of REALIST ORBCEL-C cells on:

1. Physiological indices of respiratory dysfunction reflecting severity of ARDS, as measured by oxygenation index (OI), respiratory compliance, and P/F ratio.
2. Sequential organ failure assessment (SOFA) score.
3. Extubation and reintubation
4. Ventilation free days at day 28
5. Duration of ventilation
6. Length of ICU and hospital stay
7. 28-day and 90-day mortality

Population:

Patients will be prospectively screened daily. All patients with moderate to severe ARDS will be entered into a screening log. If possible during the phase 2 trial, all patients with moderate to severe ARDS due to COVID-19 or other causes of ARDS will be entered into a screening log. If the patient is not recruited the reason will be recorded. A fully anonymised minimal dataset will be recorded on these patients (age, gender, APACHE II score, worst P/F ratio at time of assessment, reasons for non-enrolment and vital status). APACHE II score and vital status will be collected using anonymised linkage to the ICNARC database through a defined CMP number (or equivalent). This will allow comparison to identify that the study population is representative of the overall cohort of patients. This information is required to establish an unbiased study population and to ensure the study can be reported in keeping with CONSORT guidelines (www.consort-statement.org).

Patient consent:

Informed consent procedure:

The study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki. The chief investigator (CI) (or designee) is responsible for ensuring that informed consent for trial participation is given by each patient or a legal representative. An appropriately trained doctor or nurse may take consent. The person taking informed consent must be GCP trained, suitably qualified and experienced and have been delegated this duty on the delegation log. Appropriate signatures and dates must be obtained on the informed consent documentation prior to collection of trial data and administration of the trial drug. If no consent is given a patient cannot be randomised into the trial. The incapacitating nature of the condition precludes obtaining prospective informed consent from participants. In this situation informed consent will be sought from a Personal Legal Representative or Professional Legal representative.

Personal legal representative consent:

Informed consent will be sought from the patient's personal legal representative (Per LR) who may be a relative, partner or close friend. The Per LR will be informed about the trial by the responsible clinician or a member of the research team and provided with a copy of the covering statement for the Per LR with an attached participant information sheet (PIS) and asked to give an opinion as to whether the patient would object to taking part in such medical research. If the Per LR decides that the patient would have no objection to participating in the trial the Per LR will be asked to sign the Per LR consent form which will then be countersigned by the person taking consent. The original will be retained in the trial site file and a copy given to the Per LR and another copy placed in the patients' medical records.

During the COVID-19 pandemic, there are likely to be visiting restrictions in place due to infection control measures and therefore it may not be possible to obtain consent from the PerLR at the clinical site. If the PerLR is not available at the site, the research may contact the PerLR by telephone and seek verbal agreement. The verbal agreement will be recorded in the PerLR Telephone Agreement Form.

Professional legal representative consent:

As the patient is unable to give informed consent and no Per LR is available, a doctor who is not connected with the conduct of the trial may act as a professional legal representative (Prof LR). The doctor will be informed about the trial by the responsible clinician or a member of the research team and given a copy of the PIS. If the doctor decides that the patient is suitable for entry into the trial that doctor will be asked to sign the professional legal representative consent form. The original will be retained in the trial site file and a copy given to the Prof LR and another copy placed in the patients' medical records.

Retrospective patient consent:

Patients will be informed of their participation in the trial by the responsible clinician or a member of the research team once the patient regain capacity to understand the details of the trial. The responsible clinician or a member of the research team will discuss the study with the patient and the patient will be given a copy of the PIS to keep. The patient will be asked for consent to participate in the trial and to sign the consent to continue form which will then be countersigned by the person taking consent. The original will be retained in the trial site file and a copy given to the patient and another copy placed in the patients' medical records. Where consent to continue is not obtained, consent from the legal representative will remain valid. If the patient refuses consent, permission to use data collected to that point and to access medical records for trial data will be requested from the patient.

Withdrawal of consent:

Patients may withdraw or be withdrawn (by Per LR or Prof LR) from the trial at any time without prejudice.

In the event of a request to withdraw from the study, the researcher will determine which elements of the trial are to be withdrawn from the following possibilities and this will be documented:

* Orbcel-C administration if ongoing
* On-going data collection during hospital admission
* Confirmation of vital status
* On-going data collection following hospital discharge In the event that the request is to withdraw from all elements of the study, only anonymised data recorded up to the point of withdrawal will be included in the study analysis.

Consent will also be requested to use the samples collected to that point.

Investigational medicinal product

The Investigational Medicinal Products are:

1. Allogeneic donor CD362 enriched human umbilical cord-derived mesenchymal stromal cells (REALIST ORBCEL-C) supplied as a sterile, single-use cryopreserved cell suspension containing a fixed cell dose of either 100 x 10^6, 200 x 10^6 or 400 x 10^6 cells in 10mL, 20mL or 40mL volumes, respectively to be further diluted in Plasma-Lyte 148 to a total volume of 200mls for the purposes of administration.
2. Plasma-Lyte 148 Solution for Infusion (200mls) as the placebo control solution.

Storage, thawing and reconstitution of Orbcel-C cells:

Trial guidelines will provide detailed information regarding the protocol for storage, thawing and reconstitution, and administration of the cell product Orbcel-C and placebo.

Drug storage:

The study drug will be commenced as soon as possible following reconstitution and within 6 hours.

Study drug termination criteria:

Study drug will be continued until one of the following is met:

1. Study drug related adverse event
2. Death or discontinuation of active treatment
3. Request from Per LR or Pro LR to withdraw the patient from the study
4. Decision by the attending clinician on safety grounds.

Study drug compliance:

Any omission of the study drug will be recorded in the CRF to monitor compliance.

Study drug accountability:

The site clinical trials pharmacist and cell therapy facility staff will maintain full accountability for the study drug received, prepared and dispensed to patients in ICU. Records will be kept allowing traceability between the cell donor and the IMP recipient. Drug administration will be recorded on the patient's prescription chart.

Study drug return and destruction:

Any partially used study drug should be disposed of/destroyed at the site in accordance with Trial guidelines and local biological waste management policies.

Unused product should disposed of/destroyed under the supervision of the site clinical trials pharmacist. Records of return and destruction will be maintained.

Data Quality:

The NICTU will provide training to site staff on trial processes and procedures including CRF completion and data collection. Within the NICTU the clinical data management process is governed by SOPs to ensure standardisation and adherence to International Conference on Harmonisation Good Clinical Practice (ICH GCP) guidelines and regulatory requirements. Data is to be entered onto the electronic database as per the CRF entry timelines. On-site monitoring visits during the trial will check: (i) the accuracy of the data entered into the CRF, (ii) entries against source documents alongside adherence to the protocol, (iii) trial specific procedures and (iv) Good Clinical Practice (GCP). This monitoring will be carried out as per the trial specific Monitoring Plan. Changes to data will be recorded and fully auditable. Data errors will be documented and corrective actions implemented. Data validation will be implemented and discrepancy reports will be generated following data entry to identify data that may be out of range or inconsistent, or protocol deviations, based on data validation checks programmed into the clinical trial database. For routinely collected clinical data the NHS record will be the source document and for study specific measurements the CRF will be the source document.

Data management:

The PI (or designee) will collect all data and record this in the CRF. Each participant will be allocated a unique participant study number at trial entry, and this, and initials, will be used to identify him or her on the CRF for the duration of the trial. Data will be collected from the time of trial entry until hospital discharge. Trial data will be entered onto a CRF and processed electronically as per NICTU SOPs and the study specific Data Management Plan (DMP). Submitted data will be reviewed for completeness and entered onto a secure, backed-up custom database. Due care will be taken to ensure data safety and integrity, and compliance with GDPR and the Data Protection Act 2018. Data queries will be raised electronically. The designated site staff will be required to respond to these queries within 2 weeks and send them back to the CTU after the queries have been reviewed and signed by the CI/delegated staff member. Any amended information will then be entered in the study database. A copy of the signed data query form should be retained with the CRF at the investigator site.

If the participant is transferred to another hospital the PI or designated member of the site study team will liaise with the receiving hospital to ensure complete data capture as per CRF instruction. If this is not possible, the primary outcome must be collected as a minimum. CRFs are to be submitted to the CTU as per the CRF submission schedule. Data censorship for each trial will occur 90 days post randomisation.

Analysis Population The primary analysis will be conducted on all outcome data obtained from all participants regardless of protocol adherence, i.e. intention to treat analysis.

It is possible that some enrolled subjects may not be treated with study drug. Therefore a secondary analysis of the all-treated population analysis will be undertaken.

For the Phase 1 trial no formal statistical analysis will be performed on safety data. The primary analysis will be descriptive and will focus on adverse events. The number of pre specified cell infusion associated events will also be reported. Descriptive analysis of pulmonary and non-pulmonary organ function will also be undertaken. We plan to publish the data from the phase 1 study.

In the completed Phase 1 REALIST trial, infusion of 400 million cells was achieved without any dose limiting toxicity at day 7 and has been approved by the DMEC as the intervention dose for this study.

For the Phase 2 trial, adverse events will be reported as for the Phase 1 study. For continuously distributed outcomes, differences between groups will be tested using independent samples t-tests and analysis of covariance with transformations of variables to normality if appropriate, or non-parametric equivalents. Chi-square tests (or Fisher's Exact tests) will be used for categorical variables. A p value of 0.05 will be considered as significant.

Correlations between changes in the biological markers measured and physiological and clinical outcomes will be assessed by appropriate graphical and statistical methods including Pearson's (or Spearman's) correlation coefficient.

A final analysis and report of the Phase 1 study is planned following the last patient's 90 day follow up. A final analysis and report of the phase 2 study is planned following the last patient's 90 day follow up. The 2 year follow up data will be published thereafter and will be an important long term outcome. A detailed statistical analysis plan will be written and approved by the independent DMEC prior to any analysis.

All the power calculations and methodology for data analysis have been confirmed by the trial statistician from the Northern Ireland Clinical Trials Unit (NICTU).

Missing data:

Every effort will be made to minimise missing baseline and outcome data in this trial. The level and pattern of the missing data in the baseline variables and outcomes will be established by forming appropriate tables and the likely causes of any missing data will be investigated. This information will be used to determine whether the level and type of missing data has the potential to introduce bias into the analysis results for the proposed statistical methods, or substantially reduce the precision of estimates related to treatment effects. If necessary, these issues will be dealt with using multiple imputation or Bayesian methods for missing data as appropriate.

Sample size:

The phase 1 trial will recruit up to 18 participants. The sample size for the phase 2 REALIST trial is 60 patients with ARDS due to COVID-19 and 60 patients with ARDS not due to COVID-19 (30 in each of the ORBCEL-C and placebo groups). Due to the clinical differences in patients with ARDS due to COVID-19 and other causes of ARDS, patients with ARDS due to COVID-19 and other causes of ARDS will be recruited as separate cohorts. This will also facilitate timely reporting of the results from each cohort.

Although the primary focus of the phase 2 trial is safety, there is, however, power to detect a difference in physiological outcomes.

The primary efficacy outcome measure will be the difference in oxygenation index (OI) between the ORBCEL-C and placebo treated groups at day 7. Based on our data from a recently completed clinical trial in ARDS, the mean (standard deviation; SD) OI at day 7 in patients with ARDS is 62(51)cmH2O/kPa [4]. To allow 1:1 recruitment (ORBCEL-C vs placebo) a sample size of 56 subjects will have 80% power at a two-tailed significance level of 0.05 using a two-sample t-test to detect a clinically significant difference of 39 cmH2O/kPa in OI between groups. In a previous phase 2 study of similar size, we have found that an intervention can demonstrate a change in OI of a similar magnitude confirming a treatment effect of this size can be achieved [4].

Although we anticipate few withdrawals or loss to follow-up we have allowed for this in the sample size calculation. In previous UK multicentre studies in the critically ill <3% withdrew consent or were lost to follow-up [4, 65]. Therefore, a conservative drop-out rate of 5% has been estimated and the study will require a total of 60 patients (30 patients in the ORBCEL-C and 30 in the placebo group).

ELIGIBILITY:
Inclusion Criteria:

1. ARDS as defined by the Berlin definition.

   1. Onset within 1 week of identified insult.
   2. Within the same 24-hour time period i. Hypoxic respiratory failure (PaO2/ FiO2 ratio ≤ 27kPa on PEEP ≥ 5 cmH20) ii. Bilateral infiltrates on chest X-ray consistent with pulmonary oedema not explained by another pulmonary pathology iii. Respiratory failure not fully explained by cardiac failure or fluid overload
2. Patient is receiving invasive mechanical ventilation
3. COVID-19 based on clinical diagnosis or PCR result or other causes of ARDS.

Exclusion Criteria:

1. More than 72 hours from the onset of ARDS.
2. Age < 16 years.
3. Patient is known to be pregnant
4. Major trauma in the prior 3 days.
5. Presence of any active malignancy (other than non-melanoma skin cancer) that required treatment within the last year.
6. WHO Class III or IV pulmonary hypertension.
7. Venous thromboembolism currently receiving anti-coagulation or within the past 3 months
8. Currently receiving extracorporeal life support (ECLS).
9. Severe chronic liver disease with Child-Pugh score > 12.
10. DNAR (Do Not Attempt Resuscitation) order (excluding advance directives) in place.
11. Treatment withdrawal imminent within 24 hours.
12. Consent declined.
13. Prisoners.
14. Non-English speaking patients or those who do not adequately understand verbal or written information unless an interpreter is available.
15. Previously enrolled in the REALIST trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Oxygenation index (OI) | Day 7
  OI is a physiological index of the severity of ARDS and measures both impaired oxygenation and the amount of mechanical ventilation delivered
Incidence of Serious Adverse Events (SAEs) | 90 days
  Incidence of SAEs

SECONDARY OUTCOMES:
Oxygenation index | Days 4 and 14
Sequential Organ Failure Assessment (SOFA) score | Days 4, 7 and 14
  SOFA score is a measure of organ failure
Respiratory compliance (Crs) | Days 4, 7 and 14
  Crs is a physiological measure of pulmonary function in ARDS
Partial pressure of arterial oxygen to the fraction of inspired oxygen ratio (P/F ratio) | Days 4, 7 and 14
  P/F ratio is a physiological measure of pulmonary function in ARDS
Driving Pressure | Days 4, 7 and 14
Extubation and reintubation | Up to day 14 or until the patient is discharged from ICU or the patient dies
Ventilation free days at day 28 | Day 28
Length of ICU and hospital stay | Until the patient is discharged or the patient dies
28-day and 90-day mortality | Up to 28 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Danny F McAuley, Professor, Principal Investigator — Belfast Health and Social Care Trust
Locations (1):
- Belfast Health and Social Care Trust, Royal Hospitals, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gorman EA, Rynne J, Gardiner HJ, Rostron AJ, Bannard-Smith J, Bentley AM, Brealey D, Campbell C, Curley G, Clarke M, Dushianthan A, Hopkins P, Jackson C, Kefela K, Krasnodembskaya A, Laffey JG, McDowell C, McFarland M, McFerran J, McGuigan P, Perkins GD, Silversides J, Smythe J, Thompson J, Tunnicliffe WS, Welters IDM, Amado-Rodriguez L, Albaiceta G, Williams B, Shankar-Hari M, McAuley DF, O'Kane CM. Repair of Acute Respiratory Distress Syndrome in COVID-19 by Stromal Cells (REALIST-COVID Trial): A Multicenter, Randomized, Controlled Clinical Trial. Am J Respir Crit Care Med. 2023 Aug 1;208(3):256-269. doi: 10.1164/rccm.202302-0297OC. PMID 37154608
- [Derived] Gorman E, Shankar-Hari M, Hopkins P, Tunnicliffe WS, Perkins GD, Silversides J, McGuigan P, Jackson C, Boyle R, McFerran J, McDowell C, Campbell C, McFarland M, Smythe J, Thompson J, Williams B, Curley G, Laffey JG, Clarke M, McAuley DF, O'Kane C. Repair of acute respiratory distress syndrome by stromal cell administration (REALIST): a structured study protocol for an open-label dose-escalation phase 1 trial followed by a randomised, triple-blind, allocation concealed, placebo-controlled phase 2 trial. Trials. 2022 May 13;23(1):401. doi: 10.1186/s13063-022-06220-0. PMID 35562778
- [Derived] Gorman E, Shankar-Hari M, Hopkins P, Tunnicliffe WS, Perkins GD, Silversides J, McGuigan P, Krasnodembskaya A, Jackson C, Boyle R, McFerran J, McDowell C, Campbell C, McFarland M, Smythe J, Thompson J, Williams B, Curley G, Laffey JG, Clarke M, McAuley DF, O'Kane CM. Repair of acute respiratory distress syndrome by stromal cell administration (REALIST) trial: A phase 1 trial. EClinicalMedicine. 2021 Oct 24;41:101167. doi: 10.1016/j.eclinm.2021.101167. eCollection 2021 Nov. PMID 34746723
- [Derived] Gorman E, Shankar-Hari M, Hopkins P, Tunnicliffe WS, Perkins GD, Silversides J, McGuigan P, Jackson C, Boyle R, McFerran J, McDowell C, Campbell C, McFarland M, Smythe J, Thompson J, Williams B, Curley G, Laffey JG, Clarke M, O'Kane C, McAuley DF. Repair of Acute Respiratory Distress Syndrome by Stromal Cell Administration in COVID-19 (REALIST-COVID-19): A structured summary of a study protocol for a randomised, controlled trial. Trials. 2020 Jun 3;21(1):462. doi: 10.1186/s13063-020-04416-w. PMID 32493473